CLINICAL TRIAL: NCT00983918
Title: Postoperative Pain After Laparoscopic Cholecystectomy After Anesthesia With Isoflurane, Desflurane, Sevoflurane or Propofol
Brief Title: Pain After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Jaime Ortiz, Assistant Professor of Anesthesiology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-24815
Record Dates: First submitted 2009-09-22; First posted 2009-09-24 (Estimated); Results first posted 2014-03-11 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Desflurane; Sevoflurane; Isoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Desflurane (Active Comparator): General Anesthesia with Desflurane
  Interventions: Drug: Desflurane
- Sevoflurane (Active Comparator): General Anesthesia with Sevoflurane
  Interventions: Drug: Sevoflurane
- Isoflurane (Active Comparator): General Anesthesia with Isoflurane
  Interventions: Drug: Isoflurane
- Propofol (Active Comparator): General Anesthesia with Propofol
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Desflurane — Patient induced for general anesthesia as per standard protocol and maintenance of anesthesia provided with Desflurane
  Arms: Desflurane
Drug: Sevoflurane — Patient induced for general anesthesia as per standard protocol and maintenance of anesthesia provided with Sevoflurane
  Arms: Sevoflurane
Drug: Isoflurane — Patient induced for general anesthesia as per standard protocol and maintenance of anesthesia provided with Isoflurane
  Arms: Isoflurane
Drug: Propofol — Patient induced for general anesthesia as per standard protocol and maintenance of anesthesia provided with intravenous Propofol infusion
  Arms: Propofol

SUMMARY:
To the investigators' knowledge, no study has looked at differences in postoperative pain when comparing maintenance of anesthesia with isoflurane, desflurane, sevoflurane, and propofol in laparoscopic cholecystectomy. The investigators' hypothesis is that total intravenous anesthesia with propofol will lead to less postoperative pain in the first 24 hours after laparoscopic cholecystectomy when compared to maintenance of anesthesia with isoflurane, desflurane or sevoflurane.

PURPOSE

To find out if maintenance of anesthesia with propofol leads to less postoperative pain after laparoscopic cholecystectomy when compared to maintenance of anesthesia with isoflurane, desflurane, or sevoflurane.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ages 18-64
2. American Society of Anesthesiology Physical Status I, II or III
3. Inpatients scheduled to undergo laparoscopic cholecystectomy at Ben Taub General Hospital

Exclusion Criteria:

1. Open cholecystectomy - excluded due to increased levels of pain in open procedures
2. Scheduled for ambulatory surgery
3. Renal dysfunction (Serum Cr > 1.2) - excluded due to potential altered metabolism of anesthetic and pain medications
4. Allergy to any of the study medications or anesthetic agents
5. Chronic opioid analgesic use at home - excluded due to potential difficulty in assessing pain caused by the procedure alone
6. Patient inability to properly describe postoperative pain to investigators (language barrier, dementia, delirium, psychiatric disorder)
7. Patient or surgeon refusal

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Ortiz, MD, Principal Investigator — Baylor College of Medicine, Dept. of Anesthesiology
Locations (1):
- Ben Taub General Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from September 23, 2009 to March 9, 2010/
Period: Overall Study
Arm/Group | Desflurane | Sevoflurane | Isoflurane | Propofol
Started | 20 | 20 | 20 | 20
Completed | 20 | 18 | 18 | 18
Not Completed | 0 | 2 | 2 | 2
Not completed — conversion to open cholecystectomy | 0 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desflurane | Sevoflurane | Isoflurane | Propofol | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 20 | 80
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (12) | 34 (14) | 34 (12) | 29 (7) | 33 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 16 | 18 | 63
  Male | 6 | 5 | 4 | 2 | 17
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 20 | 80

OUTCOME MEASURES:

1. Primary Outcome: Pain Measured on Verbal Scale of 0-10
Description: Pain measured on verbal scale of 0-10, with 0 being absolutely no pain, and 10 being the worst pain in that subjects life.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Desflurane | Sevoflurane | Isoflurane | Propofol
Number analyzed (Participants) | 20 | 18 | 18 | 18
units on a scale | 2.7 (3.2) | 1.7 (2.4) | 3 (2.5) | 2.1 (1.4)

ADVERSE EVENTS:
Arm/Group | Desflurane | Sevoflurane | Isoflurane | Propofol
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/20 | 0/18 | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes